CLINICAL TRIAL: NCT00317993
Title: Effects of Ezetimibe and Simvastatin on LDL Receptor Protein Expression and on LDL Receptor and HMG-CoA Reductase mRNA Expression in Mononuclear Cells: a Randomized Controlled Study in Healthy Men
Brief Title: LDL Receptor Under Ezetimibe and Simvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EZE04-003
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Men
MeSH Terms: interventions — Ezetimibe; Simvastatin

INTERVENTIONS:
Drug: ezetimibe
Drug: simvastatin
Drug: ezetimibe plus simvastatin

SUMMARY:
The purpose of this study is to investigate the effects of the two lipid -lowering drugs, ezetimibe and simvastatin, on lipid metabolism in humans. In specific, the study will investigate in blood cells whether the enzyme that controls cholesterol synthesis, HMG-CoA reductase, and the receptor that takes up cholesterol from the blood, the LDL receptor, are changed during treatment with the aforementioned drugs.

DETAILED DESCRIPTION:
Ezetimibe decreases serum total and LDL cholesterol levels by blocking cholesterol absorption in the intestine, causing a compensatory increase in cholesterol synthesis. The exact underlying regulatory mechanisms of the ezetimibe-induced increase in cholesterol synthesis and decrease in serum LDL cholesterol are not known. In addition, it has never been investigated whether changes in LDL receptor expression contribute to the LDL-lowering effect of ezetimibe, as is the case with other agents causing a decrease in cholesterol absorption such as the plant stanols.

In the present study, we plan to examine changes in LDL receptor and HMG-CoA reductase mRNA concentrations during ezetimibe treatment. For comparison, effects of simvastatin and the combined administration of the two will be investigated. Since mRNA expression profiles provide information about effects at the transcriptional but not necessarily at the translational level, we will also analyze changes in the LDL receptor protein at the cell surface of mononuclear blood cells. As a functional marker for HMG-CoA reductase activity the ratio of serum lathosterol to cholesterol concentration will be used since it correlates with HMG-CoA reductase activity and serves also as a marker of total cholesterol synthesis.

In this regard it has been shown that plant sterols, which also act by blocking intestinal cholesterol absorption, increase cholesterol synthesis, decrease LDL synthesis, increase LDL receptor mRNA levels as well as LDL receptor protein concentrations but have no significant effect on HMG-CoA reductase expression or activity in peripheral blood mononuclear cells. Aim of this prospective ran-domized parallel study is to examine changes in HMG-CoA reductase activity/expression and in LDL receptor expression/protein concentration in mononuclear blood cells under treatment with ezetimibe.

For this purpose 3 parallel groups of 20 healthy men will be formed. One group will be treated with ezetimibe (10 mg/day), one with 40 mg/day of simvastatin and another with ezetimibe (10 mg/day) plus simvastatin (40 mg/day). Each treatment period will last for 2 weeks. Blood drawing will be per-formed at baseline (before the initiation of treatment) and at the end of the 2 weeks. (storing of the samples at -80°). The measurements involved in this study include the determination of the lipopro-tein concentrations in serum, isolation of the mononuclear cells, measurement of LDL receptor mRNA from the peripheral blood mononuclear cells, measurement of HMG-CoA reductase mRNA levels in peripheral blood mononuclear cells, measurement of the LDL-receptor protein concentrations on the surface of peripheral blood mononuclear cells. Furthermore, the serum latosterol to cholesterol con-centrations will be measured as a surrogate marker of the HMG-CoA reductase activity.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* age between 18 and 60 years
* body mass index between 18.5 and 30 kg/m2
* LDL cholesterol smaller than 190 mg/dL
* triglicerides smaller than 250 mg/dL
* normal blood pressure

Exclusion Criteria:

* intake of lipid-lowering drugs
* excessive alcohol intake
* liver disease
* kidney disease
* coronary heart disease
* eating disorders
* diabetes or other endocrine disorders
* medications that interfere with lipid metabolism

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2004-04; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
HMG-CoA reductase activity
HMG-CoA reductase mRNA expression
LDL receptor mRNA expression
LDL receptor protein

CONTACTS AND LOCATIONS:
Overall Officials: Ioanna Gouni-Berthold, MD, Principal Investigator — Medizinische Klinik II und Poliklinik für Innere Medizin
Locations (1):
- Medizinische Klinik II und Poliklinik für Innere Medizin, Cologne, Germany

REFERENCES:
- [Derived] Berthold HK, Rizzo M, Spenrath N, Montalto G, Krone W, Gouni-Berthold I. Effects of lipid-lowering drugs on high-density lipoprotein subclasses in healthy men-a randomized trial. PLoS One. 2014 Mar 24;9(3):e91565. doi: 10.1371/journal.pone.0091565. eCollection 2014. PMID 24662777
- [Derived] Gouni-Berthold I, Berthold HK, Huh JY, Berman R, Spenrath N, Krone W, Mantzoros CS. Effects of lipid-lowering drugs on irisin in human subjects in vivo and in human skeletal muscle cells ex vivo. PLoS One. 2013 Sep 2;8(9):e72858. doi: 10.1371/journal.pone.0072858. eCollection 2013. PMID 24023786
- [Derived] Berthold HK, Seidah NG, Benjannet S, Gouni-Berthold I. Evidence from a randomized trial that simvastatin, but not ezetimibe, upregulates circulating PCSK9 levels. PLoS One. 2013;8(3):e60095. doi: 10.1371/journal.pone.0060095. Epub 2013 Mar 27. PMID 23544125
- [Derived] Berthold HK, Berneis K, Mantzoros CS, Krone W, Gouni-Berthold I. Effects of simvastatin and ezetimibe on interleukin-6 and high-sensitivity C-reactive protein. Scand Cardiovasc J Suppl. 2013 Feb;47(1):20-7. doi: 10.3109/14017431.2012.734635. Epub 2012 Oct 18. PMID 23013513
- [Derived] Berneis K, Rizzo M, Berthold HK, Spinas GA, Krone W, Gouni-Berthold I. Ezetimibe alone or in combination with simvastatin increases small dense low-density lipoproteins in healthy men: a randomized trial. Eur Heart J. 2010 Jul;31(13):1633-9. doi: 10.1093/eurheartj/ehq181. Epub 2010 Jun 6. PMID 20525999